CLINICAL TRIAL: NCT02575833
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of AMG 334 on Exercise Time During a Treadmill Test in Subjects With Stable Angina
Brief Title: Treadmill Cardiovascular Safety Study of Erenumab (AMG 334)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140254; 2015-002322-40 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-15 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Stable Angina
Keywords: Angina; Stable Angina; Cardiovascular Disease; Exercise-induced Angina
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Cardiovascular Diseases | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single dose of placebo administered by intravenous infusion on day 1.
  Interventions: Drug: Placebo
- Erenumab (Experimental): Participants received a single dose of erenumab 140 mg administered by intravenous infusion on day 1.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — A single dose of erenumab 140 mg infused over approximately 60 minutes.
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab
Drug: Placebo — A single dose of a matching volume of placebo infused over approximately 60 minutes.
  Arms: Placebo

SUMMARY:
A phase 2a, multicenter, randomized, double-blind, placebo-controlled study in adults with stable angina to evaluate the effect of erenumab (AMG 334) compared to placebo on exercise time during an exercise treadmill test.

ELIGIBILITY:
Inclusion Criteria

* History of chronic stable angina or at least 3 months prior to screening, with at least 1 angina episode per month
* Ischemic heart disease documented by myocardial infarction, coronary angiography or a revascularization procedure
* Receiving stable doses of cardiac medication
* Completes 2 exercise treadmill tests during screening meeting protocol requirements

Exclusion Criteria:

* Participating in another investigational study
* Current or prior malignancy within 5 years of randomization
* Known sensitivity to any components of the investigational product
* Not able to complete all protocol required study visits
* Having the following within 3 months prior to or during screening: Unstable angina or acute coronary syndrome, transient Ischemic attack (TIA) or stroke, revascularization procedure, or instability in ST-segment depression between screening exercise treadmill tests, as assessed by the core electrocardiograph (ECG) laboratory

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (8):
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Las Vegas, Nevada
  - Research Site, Jackson, Tennessee
  - Research Site, New Braunfels, Texas
  - Research Site, Wichita Falls, Texas
- Bulgaria (2):
  - Research Site, Haskovo
  - Research Site, Sofia
- Czechia (4):
  - Research Site, Brandýs nad Labem
  - Research Site, Chomutov
  - Research Site, Prague
  - Research Site, Pribram VIII
- Research Site, Riga, Latvia
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Zabrze
- Research Site, Timișoara, Romania
- Slovakia (8):
  - Research Site, Bardejov
  - Research Site, Brezno
  - Research Site, Lučenec
  - Research Site, Piešťany
  - Research Site, Prešov
  - Research Site, Svidník
  - Research Site, Trenčín
  - Research Site, Žilina
- Research Site, Parow, Western Cape, South Africa
- Research Site, Geneva, Switzerland

REFERENCES:
- [Background] Depre C, Antalik L, Starling A, Koren M, Eisele O, Lenz RA, Mikol DD. A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Erenumab on Exercise Time During a Treadmill Test in Patients With Stable Angina. Headache. 2018 May;58(5):715-723. doi: 10.1111/head.13316. PMID 29878340
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 centers across the United States, South Africa, New Zealand, and the European Union (EU). Participants were enrolled from November 2015 to January 2017.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either a single dose of erenumab 140 mg or placebo intravenously (IV) prior to starting an exercise treadmill test. Randomization was stratified by the total exercise time average (< 7 minutes or ≥ 7 minutes) of the 2 qualifying exercise treadmill tests performed during screening.
Groups:
- Placebo: Participants randomized to receive a single dose of placebo administered by intravenous infusion on day 1 prior to starting an exercise treadmill test.
- Erenumab: Participants randomized to receive a single dose of erenumab 140 mg administered by intravenous infusion on day 1 prior to starting an exercise treadmill test.
Period: Overall Study
Arm/Group | Placebo | Erenumab
Started | 44 | 45
Received Study Drug | 44 | 44
Completed | 43 | 44
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.6) | 61.8 (10.1) | 62.6 (9.9)
Age, Customized [Count of Participants; unit: Participants]
  18 - < 65 years | 21 | 23 | 44
  65 - 85 years | 23 | 22 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 33 | 36 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 42 | 44 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Black (or African American) | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 37 | 43 | 80
  Multiple | 0 | 0 | 0
  Other | 2 | 0 | 2
Baseline Total Exercise Time [Mean (Standard Deviation); unit: seconds] — Total exercise time (TET) was assessed using an exercise treadmill test according to the standard Bruce protocol.
  The Bruce protocol is a standardized multistage treadmill test for assessing cardiovascular health, where the participant walks on an uphill treadmill in a graded exercise test with electrodes on the chest to monitor cardiac function. Every 3 minutes, the speed and incline of the treadmill are increased. There are 7 such stages for a total possible exercise time of 21 minutes. Population: Participants with non-missing values; baseline TET value was not calculated for two participants in the Erenumab arm due to disqualified screening values.
  seconds
    number analyzed (Participants) | 44 | 43 | 87
    (all) | 474.8 (149.5) | 490.7 (149.7) | 482.7 (148.9)
Stratification Factor: Total Exercise Time [Count of Participants; unit: Participants] — Population: Two participants in the Erenumab arm were incorrectly stratified to the < 7 minutes stratum due to disqualified screening TET values.
  Participants
    < 7 minutes | 18 | 18 | 36
    ≥ 7 minutes | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Exercise Time
Description: Total exercise time was assessed using an exercise treadmill test according to the standard Bruce protocol.
  The Bruce protocol is a standardized multistage treadmill test for assessing cardiovascular health, where the participant walks on an uphill treadmill in a graded exercise test with electrodes on the chest to monitor cardiac function. Every 3 minutes, the speed and incline of the treadmill are increased. There are 7 such stages for a total possible exercise time of 21 minutes.
Time Frame: Baseline and day 1, after dosing
Population: Participants who received study drug and completed the baseline and post-randomization exercise treadmill tests
Measure: Least Squares Mean (Standard Error); unit: seconds
Groups:
- Placebo: Participants received a single dose of placebo administered by intravenous infusion on day 1 prior to starting an exercise treadmill test.
- Erenumab: Participants received a single dose of erenumab 140 mg administered by intravenous infusion on day 1 prior to starting an exercise treadmill test.
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 44 | 42
seconds | 8.1 (14.4) | -2.9 (14.8)
Statistical Analysis 1: Comparison: Placebo vs Erenumab; The primary endpoint was analyzed using an analysis of variance model with terms for treatment group and randomization strata (< 7 or ≥ 7 minutes). If the lower bound of the 90% confidence interval (CI) of the difference in change from baseline in exercise duration was above the non-inferiority margin of -90 seconds, then the hypothesis that erenumab does not decrease exercise duration would be supported; Test type: Non-Inferiority — The non-inferiority margin was -90 seconds; Treatment Difference = -11.0, 90% CI 2-sided [-44.9 to 22.9], Standard Error of Mean 20.4

2. Secondary Outcome: Time to Onset of Exercise-induced Angina
Description: Time to onset of angina was defined as the time the participant received study drug to the time of event onset during the exercise treadmill test. If no event occurred the participant was censored at the exercise treadmill test stop time.
Time Frame: Day 1
Population: Participants who received study drug and completed the post-randomization exercise treadmill test
Measure: Median (90% Confidence Interval); unit: seconds
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 44 | 44
seconds | 508.0 [405.0 to 572.0] | 500.0 [420.0 to 540.0]
Statistical Analysis 1: Comparison: Placebo vs Erenumab; Test type: Superiority — The log-rank test statistic was used to compare the two treatment groups at a significance level of 0.10; p = 0.69, Stratified Log Rank; Log rank test stratified by baseline total exercise time strata (< 7 minutes or ≥ 7 minutes); Normal score = 1.55 — A normal score < 0 indicates fewer than expected events for erenumab 140 mg relative to placebo and therefore a longer survival time
Statistical Analysis 2: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.69, Cox Proportional Hazard; Adjusted by stratified baseline total exercise time strata (< 7 or ≥ 7 minutes); Hazard Ratio (HR) = 1.11, 90% CI 2-sided [0.73 to 1.69] — Hazard ratio estimates were obtained from the Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a lower average event rate and a longer exercise-induced angina free survival for erenumab 140 mg relative to placebo
Statistical Analysis 3: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.44, Cox Proportional Hazard; Adjusted by continuous baseline total exercise time; Hazard Ratio (HR) = 0.81, 90% CI 2-sided [0.52 to 1.26] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.47, Cox Proportional Hazard; Adjusted by baseline total exercise time strata (< 7 or ≥ 7 minutes), age group (< 65, ≥ 65), and sex; Hazard Ratio (HR) = 0.82, 90% CI 2-sided [0.52 to 1.28] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Time to Onset of ≥ 1 mm ST-segment Depression
Description: Time to onset of ≥ 1 mm ST-segment depression was defined as the time the participant received study drug to the time of event onset during the exercise treadmill test. If no event occurred the participant was censored at the exercise treadmill test stop time.
  Heart rate and rhythm were monitored during the exercise treadmill test by electrocardiography (ECG).
Time Frame: Day 1
Population: Participants who received study drug and completed the post-randomization exercise treadmill test.
Measure: Median (90% Confidence Interval); unit: seconds
Arm/Group | Placebo | Erenumab
Number analyzed (Participants) | 44 | 44
seconds | 420.0 [409.0 to 480.0] | 407.0 [380.0 to 443.0]
Statistical Analysis 1: Comparison: Placebo vs Erenumab; Test type: Superiority — The log-rank test statistic was used to compare the two treatment groups at a significance level of 0.10; p = 0.59, Stratified Log Rank; Log rank test stratified by baseline total exercise time strata (< 7 minutes or ≥ 7 minutes); Normal score = 2.2 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.59, Cox Proportional Hazard; Adjusted by stratified baseline total exercise time strata (< 7 or ≥ 7 minutes); Hazard Ratio (HR) = 1.14, 90% CI 2-sided [0.76 to 1.69] — Hazard ratio estimates were obtained from the Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a lower average event rate and a longer exercise-induced ST-segment depression free survival for erenumab 140 mg relative to placebo
Statistical Analysis 3: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.75, Cox Proportional Hazard; Adjusted by continuous baseline total exercise time; Hazard Ratio (HR) = 1.08, 90% CI 2-sided [0.73 to 1.60] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs Erenumab; Test type: Superiority; p = 0.39, Cox Proportional Hazard; Adjusted by baseline total exercise time strata (< 7 or ≥ 7 minutes), age group (< 65, ≥ 65), and sex; Hazard Ratio (HR) = 1.24, 90% CI 2-sided [0.82 to 1.87] — [estimate comment as in outcome 3, analysis 2]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Erenumab 140 mg: Participants received a single dose of erenumab 140 mg administered by intravenous infusion on day 1 prior to starting an exercise treadmill test.
Arm/Group | Placebo | Erenumab 140 mg
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/44
Other Adverse Events (participants affected / at risk) | 6/44 | 4/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Erenumab 140 mg (N=44)
Atrial fibrillation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Erenumab 140 mg (N=44)
Influenza (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02575833/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02575833/SAP_001.pdf